CLINICAL TRIAL: NCT05147415
Title: A Phase 2b, Double-blind, Randomized, Placebo-controlled, Dose-finding, Multi-center, 36-week Safety and Efficacy Study With Open-label Extension (OLE) Period of Tesomet in Subjects With Hypothalamic Obesity
Brief Title: Study of Tesomet With Open-label Extension in Subjects With Hypothalamic Obesity (HO)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to financial considerations Sponsor is unable to complete the trial and assess the planned objectives/endpoints. No subjects have been randomized to treatment in the clinical trial and the decision therefore has no safety concern for patients
Sponsor: Saniona (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TM008
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Hypothalamic Obesity
MeSH Terms: conditions — Sexual Infantilism | interventions — Tesofensine; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Once-daily PO for 36 weeks during the double-blind period; then if continued eligible for OLE, once-daily dosing for 36 weeks at the highest tolerated Tesomet dose from the double-blind period
  Interventions: Other: Placebo; Drug: Tesomet
- Tesomet Low Dose (Experimental): Once-daily PO for 36 weeks during the double-blind period; then if continued eligible for OLE, once-daily dosing for 36 weeks at the highest tolerated dose from the double-blind period
  Interventions: Drug: Tesomet
- Tesomet Medium Dose (Experimental): Once-daily PO for 36 weeks during the double-blind period; then if continued eligible for OLE, once-daily dosing for 36 weeks at the highest tolerated dose from the double-blind period
  Interventions: Drug: Tesomet
- Tesomet High Dose (Experimental): Once-daily PO for 36 weeks during the double-blind period; then if continued eligible for OLE, once-daily dosing for 36 weeks at the highest tolerated dose from the double-blind period
  Interventions: Drug: Tesomet

INTERVENTIONS:
Other: Placebo — Inactive comparator
  Arms: Placebo
Drug: Tesomet — Fixed-dose combination
  Other Names: tesofensine; metoprolol

SUMMARY:
This study will evaluate the safety and efficacy of Tesomet (tesofensine + metoprolol) in subjects 18 years of age or older, with HO

ELIGIBILITY:
Key Inclusion Criteria:

* Subject and, if applicable, their parent or legal guardian must be willing to provide informed consent
* Diagnosis of HO secondary to damage to the hypothalamus
* Female subjects must be of non-childbearing potential
* At least 6 months since completion of therapy (chemotherapy, surgery, or radiation with resulting injury to the hypothalamus and/or the pituitary) with stable disease and lack of recurrence
* BMI 30.0 to 60.0 kg/m², inclusive
* Documented stable body weight (gain/loss <10%) for at least 90 days prior to Screening
* Stable and well-managed pituitary replacement (eg, glucocorticoid, thyroid hormone, estrogen/progestin or testosterone, desmopressin, or growth hormone) for >2 months prior to Screening
* Male subjects who are sexually active must be surgically sterile

Key Exclusion Criteria:

* Females who are pregnant, breastfeeding, or actively intending to become pregnant during the study
* Sitting BP that meets the following criteria after 5 minutes of rest at Screening:

  1. Systolic BP >145 mmHg or <100 mmHg; or
  2. Diastolic BP >95 mmHg or <70 mmHg
* Type 1 diabetes mellitus
* History of major depressive disorder within 2 years prior to Screening, or any history of other severe psychiatric disorder (eg, schizophrenia, bipolar disorder)
* Uncontrolled endocrine disorders (eg, Cushing syndrome, Addison's, hypothyroidism, hyperthyroidism)
* History of bulimia or anorexia nervosa
* Use of prohibited medications, including current use of selective serotonin reuptake inhibitors / serotonin-norepinephrine reuptake inhibitors (SSRIs/SNRIs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Body weight (%) | Baseline to Week 36
  Percentage change in body weight

SECONDARY OUTCOMES:
Body weight loss | Week 36
  Proportion of subjects who meet pre-specified thresholds for body weight loss
Body weight (kg) | Baseline to Week 36
  Change in body weight in kilograms
Waist circumference (cm) | Baseline to Week 36
  Change in waist circumference in centimeters
Body Mass Index (BMI) | Baseline to Week 36
  Change in BMI

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Guillaume, MS, Study Director — Saniona
Locations (1):
- Sparrow Clinical Research Institute, Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The Sponsor will consider requests from qualified researchers for access to TM008 study materials
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Following completion of Tesomet clinical development